CLINICAL TRIAL: NCT00453687
Title: A Single-centre, Randomized, Double-blind Placebo-controlled, Dose-ascending, Cross-over Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Inhaled Doses of GSK233705, Formulated With the Excipient Magnesium Stearate, in Healthy Volunteers
Brief Title: A Single Centre Randomized Study Evaluating The Safety And Tolerability Of GSK233705 In Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AC2108380
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; GSK233705,; Magnesium Stearate,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Drug
  Interventions: Drug: GSK233705

INTERVENTIONS:
Drug: GSK233705 — investigational drug

SUMMARY:
This study will investigate the safety and tolerability of inhaled doses of GSK233705 with a new formulation.

DETAILED DESCRIPTION:
A single-centre, randomized, double-blind placebo-controlled, dose-ascending, cross-over study to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of single inhaled doses of GSK233705 (50, 100 and 200Âµg), formulated with the excipient magnesium stearate, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 18-55 years old
* Non-Smokers

Exclusion Criteria:

* Any subject with breathing problems.
* High blood pressure and heart abnormalities.
* Any subjects currently taking prescription and non-prescription medications.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03-09 (Actual); Primary Completion 2007-05-16 (Actual); Study Completion 2007-05-16 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability endpoints: adverse events, blood pressure, heart rate, 12-lead electrocardiogram (ECG), Holter and Lead II ECG monitoring, lung function (FEV1, FVC) and clinical laboratory safety tests over 24 hours. | over 24 hours.

SECONDARY OUTCOMES:
Plasma and urine concentrations of GSK233705 and derived pharmacokinetic parameters from 0 to 24 hours. Serial Specific airway conductance (sGaw) and Forced Expiratory Volume in 1 second (FEV1) measurements over 24 hours post-dose. | over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study AC2108380 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/AC2108380?search=study&search_terms=AC2108380#rs
- Available data/document: Study Protocol: AC2108380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AC2108380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC2108380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC2108380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AC2108380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AC2108380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC2108380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register